CLINICAL TRIAL: NCT02738099
Title: Risk Stratification of Patients Presenting With Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Essentia Health (Other)
Responsible Party: Principal Investigator, Michael Mollerus, MD, Essentia Health
Other Study IDs: CardiacArrestSCAI
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arrest from presume Cardiac etiology: Comatose patients following arrest of presumed cardiac etiology arriving to receiving facility within 12 hours of event.

SUMMARY:
Method: Single center, prospective, non-randomized, unblinded case series of all patients presenting with a cardiac arrest. The proposed study will collect data on all comatose patients presenting with cardiac arrest. The primary end point is death from any cause at 30 days from admission.

Significance: Develop criteria to guide an invasive strategy for comatose patients presenting with cardiac arrest, and so avoid ineffective or even futile therapy which carry its own significant risks for patients in the future. The criteria, in turn, can serve as the basis for a prospective, randomized trial in the future.

DETAILED DESCRIPTION:
Research Design and Methods:

General Approach: This study is a prospective, non-randomized, unblinded case series of comatose patients presenting with cardiac arrest to either Essentia East (St. Mary's Medical Center or Miller-Dwan Medical Center) or Essentia West (Innovis Health).

Methods and Materials: Patients will be enrolled over a 60-month period by the PI, Sub-I, or study coordinator. The enrollment goal is 100 patients. The study will collect demographic, clinical and outcome data on comatose patients presenting with cardiac arrest only, and does not prescribe any clinical testing or therapies including PCI or hypothermia. All clinical decisions are left to the discretion of the attending providers.

Consent Process: This study will seek a waiver for informed consent as the patients, by study inclusion criteria, will not be able to provide informed consent, and this study uses a minimal risk design. In the spirit of transparency, attempts will be made to inform the patient, patient representative or family when possible of enrollment in the study within 48 hours of enrollment. The patient or appropriate patient representative identified from the EMR will be spoke to in person or by phone by the PI, sub-PI, or study coordinator.21 The patient and/or family will then have the opportunity to decline participation in the study. The conversation will be documented in the medical record by the PI, sub-PI or study coordinator.

Randomization Process: The study is a prospective, non-randomized, unblinded case series. Patient will be followed as a single cohort, and no randomization is required.

Study Endpoints:

Primary Endpoint:

• Death from any cause at 30 days from admission.

Secondary Endpoints:

* Death from any cause at 30 days from admission stratified by SCAI22 score
* Death from any cause at 30 days from admission stratified by presence or absence of PCI
* Neurological status at time of discharge using the Glasgow-Pittsburgh Cerebral-Perfusion Categories23,24

Observational and Data Collection:

Demographic and clinical data will be collected by a study investigator or study coordinator within 24 hours of admission. Potential candidates for participation will be identified by the PI, sub-PI, or study coordinator every morning by contacting the attending critical care or cardiology attending physicians every morning. Once identified, the study PI, sub-PI, or study coordinator will begin the chart review for data collection. Diagnostic and therapeutic management is left to the discretion of the attending providers. The protocol mandates no evaluation or therapies outside the usual practice of the attending providers. Baseline Demographic data will include:

Date of birth/Age Gender LVEF prior to admission Presence or absence of coronary artery disease Presence or absence of Comorbidities including COPD, diabetes, renal failure active malignancy, dementia, anemia Presence of congestive Presence of angina and CCS functional class heart failure and prior to admission NYHA functional Ethnicity class prior to admission

Baseline Clinical Variables that will be obtained include:25

Vitals signs on presentation to receiving facility including blood pressure, heart rate, respiratory rate, weight, height Witnessed or unwitnessed arrest Presence or absence of bystander CPR Resuscitation attempted by trained emergency personnel prior arrival at initial facility (receiving or transferring) Initial Rhythm prior to ROSC (for a pulseless arrest, the initial rhythm when the AED is placed) Therapies applied during resuscitation including CPR, defibrillation, medications, intubation Estimated time from initial arrest to initial ROSC Initial electrocardiogram characteristics including presence or absence of ST elevation, rhythm, corrected QT interval, QRS width Initial perfusing rhythm following resuscitation Time from arrival of medical personnel at scene of arrest to arrival at receiving facility. If the patient is brought to the receiving facility by someone other than medical personnel, then time is set to 0. Time to arrival to referral center from receiving facility. If referral center is also the receiving facility, then the time is set to 0. Time to arrival from receiving facility to intensive care unit or cath lab if the cath lab precedes the ICU Time to arrival to cath lab from the receiving facility Presence or absence of significance obstructive lesions and list of involved vessels if patient undergoes coronary angiography during hospitalization PCI performed and vessels treated if patient undergoes PCI during hospitalization Presence of absence of any ST elevation on an electrocardiogram within 24 hours of admission to referral facility Any use of mechanical support within 24 hours of admission to referral facility Any use of therapeutic cooling within 24 hours of admission to referral facility Any use of vasopressor agents within 24 hours of admission to referral facility Admission hemoglobin, creatine, and cardiac troponin, bicarbonate, pH, pO2 Glasgow Coma Score Presence or absence of cardiogenic shock within 24 hours of admission to referral facility Left Ventricular Ejection Fraction determined during the hospitalization and Closest to the time of death or discharge

During the clinical stay, pertinence clinical data will be collected including recurrent cardiac arrests, need for coronary angiography or revascularization more than 24 hours from admission, or implantation of an implantable cardioverter-defibrillator prior to discharge. Other significant clinical events will also be recorded including need for transfusion or other surgeries. A SCAI risk score22 will be calculated from the collected data by a study investigator or coordinator within 24 hours of admission. If the patient dies prior to discharge, the date and cause of death will be noted. Transfer to hospice or referral for comfort care will be recorded. If the patient is discharged alive, a Glasgow-Pittsburgh Cerebral Perfusion Category as a measurement of neurological function at time of discharge will be assessed. Disposition site (home, hospice, skilled nursing facility, or transfer to higher level of care) will be recorded. Thirty day follow-up will be performed by review of the medical record, review of public death records, or phone call as appropriate to assess vital status. If a recorded height or weight is not available within the first 24 hours, then estimations by either the staff caring for the patient or study coordinator may be used. The study will only collect data and will not include interaction with subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Presumed cardiac etiology of arrest
3. GCS ≤ 819,20
4. Initial presentation to an outside facility or to the emergency room of the receiving facility.

Exclusion Criteria:

1. Presumed non-cardiac etiology of arrest including trauma, pulmonary embolus, sepsis, respiratory failure.
2. GCS > 9
3. Transfer time from arrest to receiving facility greater than 12 hours
4. Cardiac arrest occurring after admission to either the outside facility or receiving facility.
5. Patient pronounced dead prior to arrival to the receiving facility emergency room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose patients presenting with cardiac arrest to the receiving facility within 12 hours of the event
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Death from any cause | 30 days
  Death from any cause at 30 days from admission

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Mollerus, MD, Principal Investigator — Essentia Health
Locations (1):
- St. Mary's MedicalCenter, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Davies MJ, Thomas A. Thrombosis and acute coronary-artery lesions in sudden cardiac ischemic death. N Engl J Med. 1984 May 3;310(18):1137-40. doi: 10.1056/NEJM198405033101801. PMID 6709008
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] Idris AH, Guffey D, Aufderheide TP, Brown S, Morrison LJ, Nichols P, Powell J, Daya M, Bigham BL, Atkins DL, Berg R, Davis D, Stiell I, Sopko G, Nichol G; Resuscitation Outcomes Consortium (ROC) Investigators. Relationship between chest compression rates and outcomes from cardiac arrest. Circulation. 2012 Jun 19;125(24):3004-12. doi: 10.1161/CIRCULATIONAHA.111.059535. Epub 2012 May 23. PMID 22623717
- [Background] Spaite DW, Bobrow BJ, Stolz U, Berg RA, Sanders AB, Kern KB, Chikani V, Humble W, Mullins T, Stapczynski JS, Ewy GA; Arizona Cardiac Receiving Center Consortium. Statewide regionalization of postarrest care for out-of-hospital cardiac arrest: association with survival and neurologic outcome. Ann Emerg Med. 2014 Nov;64(5):496-506.e1. doi: 10.1016/j.annemergmed.2014.05.028. Epub 2014 Jul 23. PMID 25064741
- [Background] Mooney MR, Unger BT, Boland LL, Burke MN, Kebed KY, Graham KJ, Henry TD, Katsiyiannis WT, Satterlee PA, Sendelbach S, Hodges JS, Parham WM. Therapeutic hypothermia after out-of-hospital cardiac arrest: evaluation of a regional system to increase access to cooling. Circulation. 2011 Jul 12;124(2):206-14. doi: 10.1161/CIRCULATIONAHA.110.986257. PMID 21747066
- [Background] Komatsu T, Kinoshita K, Sakurai A, Moriya T, Yamaguchi J, Sugita A, Kogawa R, Tanjoh K. Shorter time until return of spontaneous circulation is the only independent factor for a good neurological outcome in patients with postcardiac arrest syndrome. Emerg Med J. 2014 Jul;31(7):549-555. doi: 10.1136/emermed-2013-202457. Epub 2013 May 2. PMID 23639589
- [Background] Saravanan P, Davidson NC. Risk assessment for sudden cardiac death in dialysis patients. Circ Arrhythm Electrophysiol. 2010 Oct;3(5):553-9. doi: 10.1161/CIRCEP.110.937888. No abstract available. PMID 20959609
- [Background] Surana SP, Pun PH, Keithi-Reddy SR, Spiegel SM, Middleton JP, Singh AK. Sudden cardiac arrest in ESRD patients. Clin Nephrol. 2014 Feb;81(2):121-31. doi: 10.5414/CN107667. PMID 23149247
- [Background] Hasselqvist-Ax I, Riva G, Herlitz J, Rosenqvist M, Hollenberg J, Nordberg P, Ringh M, Jonsson M, Axelsson C, Lindqvist J, Karlsson T, Svensson L. Early cardiopulmonary resuscitation in out-of-hospital cardiac arrest. N Engl J Med. 2015 Jun 11;372(24):2307-15. doi: 10.1056/NEJMoa1405796. PMID 26061835
- [Background] Seder DB, Patel N, McPherson J, McMullan P, Kern KB, Unger B, Nanda S, Hacobian M, Kelley MB, Nielsen N, Dziodzio J, Mooney M; International Cardiac Arrest Registry (INTCAR)-Cardiology Research Group. Geriatric experience following cardiac arrest at six interventional cardiology centers in the United States 2006-2011: interplay of age, do-not-resuscitate order, and outcomes. Crit Care Med. 2014 Feb;42(2):289-95. doi: 10.1097/CCM.0b013e3182a26ec6. PMID 24107639
- [Background] Larkin GL, Copes WS, Nathanson BH, Kaye W. Pre-resuscitation factors associated with mortality in 49,130 cases of in-hospital cardiac arrest: a report from the National Registry for Cardiopulmonary Resuscitation. Resuscitation. 2010 Mar;81(3):302-11. doi: 10.1016/j.resuscitation.2009.11.021. Epub 2010 Jan 4. PMID 20047786
- [Background] Hollenbeck RD, McPherson JA, Mooney MR, Unger BT, Patel NC, McMullan PW Jr, Hsu CH, Seder DB, Kern KB. Early cardiac catheterization is associated with improved survival in comatose survivors of cardiac arrest without STEMI. Resuscitation. 2014 Jan;85(1):88-95. doi: 10.1016/j.resuscitation.2013.07.027. Epub 2013 Aug 6. PMID 23927955
- [Background] Kern KB, Lotun K, Patel N, Mooney MR, Hollenbeck RD, McPherson JA, McMullan PW, Unger B, Hsu CH, Seder DB; INTCAR-Cardiology Registry. Outcomes of Comatose Cardiac Arrest Survivors With and Without ST-Segment Elevation Myocardial Infarction: Importance of Coronary Angiography. JACC Cardiovasc Interv. 2015 Jul;8(8):1031-1040. doi: 10.1016/j.jcin.2015.02.021. Epub 2015 Jun 24. PMID 26117462
- [Background] Callaway CW, Schmicker RH, Brown SP, Albrich JM, Andrusiek DL, Aufderheide TP, Christenson J, Daya MR, Falconer D, Husa RD, Idris AH, Ornato JP, Rac VE, Rea TD, Rittenberger JC, Sears G, Stiell IG; ROC Investigators. Early coronary angiography and induced hypothermia are associated with survival and functional recovery after out-of-hospital cardiac arrest. Resuscitation. 2014 May;85(5):657-63. doi: 10.1016/j.resuscitation.2013.12.028. Epub 2014 Jan 8. PMID 24412161
- [Background] Dumas F, Cariou A, Manzo-Silberman S, Grimaldi D, Vivien B, Rosencher J, Empana JP, Carli P, Mira JP, Jouven X, Spaulding C. Immediate percutaneous coronary intervention is associated with better survival after out-of-hospital cardiac arrest: insights from the PROCAT (Parisian Region Out of hospital Cardiac ArresT) registry. Circ Cardiovasc Interv. 2010 Jun 1;3(3):200-7. doi: 10.1161/CIRCINTERVENTIONS.109.913665. Epub 2010 May 18. PMID 20484098
- [Background] Field JM, Hazinski MF, Sayre MR, Chameides L, Schexnayder SM, Hemphill R, Samson RA, Kattwinkel J, Berg RA, Bhanji F, Cave DM, Jauch EC, Kudenchuk PJ, Neumar RW, Peberdy MA, Perlman JM, Sinz E, Travers AH, Berg MD, Billi JE, Eigel B, Hickey RW, Kleinman ME, Link MS, Morrison LJ, O'Connor RE, Shuster M, Callaway CW, Cucchiara B, Ferguson JD, Rea TD, Vanden Hoek TL. Part 1: executive summary: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S640-56. doi: 10.1161/CIRCULATIONAHA.110.970889. PMID 20956217
- [Background] Rab T, Kern KB, Tamis-Holland JE, Henry TD, McDaniel M, Dickert NW, Cigarroa JE, Keadey M, Ramee S; Interventional Council, American College of Cardiology. Cardiac Arrest: A Treatment Algorithm for Emergent Invasive Cardiac Procedures in the Resuscitated Comatose Patient. J Am Coll Cardiol. 2015 Jul 7;66(1):62-73. doi: 10.1016/j.jacc.2015.05.009. PMID 26139060
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Schefold JC, Storm C, Kruger A, Ploner CJ, Hasper D. The Glasgow Coma Score is a predictor of good outcome in cardiac arrest patients treated with therapeutic hypothermia. Resuscitation. 2009 Jun;80(6):658-61. doi: 10.1016/j.resuscitation.2009.03.006. Epub 2009 Apr 11. PMID 19362767
- [Background] Passamani ER, Weisfeldt ML. 31st Bethesda Conference. Emergency Cardiac Care. Task force 3: Special aspects of research conduct in the emergency setting: Waiver of informed consent. J Am Coll Cardiol. 2000 Mar 15;35(4):862-80. No abstract available. PMID 10732882
- [Background] Brennan JM, Curtis JP, Dai D, Fitzgerald S, Khandelwal AK, Spertus JA, Rao SV, Singh M, Shaw RE, Ho KK, Krone RJ, Weintraub WS, Weaver WD, Peterson ED; National Cardiovascular Data Registry. Enhanced mortality risk prediction with a focus on high-risk percutaneous coronary intervention: results from 1,208,137 procedures in the NCDR (National Cardiovascular Data Registry). JACC Cardiovasc Interv. 2013 Aug;6(8):790-9. doi: 10.1016/j.jcin.2013.03.020. PMID 23968699
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Cummins RO, Ornato JP, Thies WH, Pepe PE. Improving survival from sudden cardiac arrest: the "chain of survival" concept. A statement for health professionals from the Advanced Cardiac Life Support Subcommittee and the Emergency Cardiac Care Committee, American Heart Association. Circulation. 1991 May;83(5):1832-47. doi: 10.1161/01.cir.83.5.1832. No abstract available. PMID 2022039